CLINICAL TRIAL: NCT01850784
Title: High Energy Formula Feeding in Infants With Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assoc Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 132/2013
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Growth Failure; Neurodevelopmental Disorder
Keywords: Congenital heart disease, Growth,Neurodevelopment
MeSH Terms: conditions — Failure to Thrive; Neurodevelopmental Disorders; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High energy formula (Active Comparator): High energy formula (Similac)
  Interventions: Dietary Supplement: High energy formula
- Standard formula (Active Comparator): Standard formula
  Interventions: Dietary Supplement: Standard formula

INTERVENTIONS:
Dietary Supplement: High energy formula — The infants with CHD will be fed with high energy formula (Similac; 1kcal/ml)
  Other Names: High energy formula (Similac)
  Arms: High energy formula
Dietary Supplement: Standard formula — The infants with CHD will be fed with standard formula (0.6-0.7 kcal/ml)
  Arms: Standard formula

SUMMARY:
High energy formula more positively affect growth in infants with congenital heart disease compared to standard formula

DETAILED DESCRIPTION:
Infants with congenital heart disease (CHD) usually show growth retardation as they can not intake enough calorie due to fluid restriction. We hypothesize that high energy formula more positively affect growth in infants with congenital heart disease compared to standard formula

ELIGIBILITY:
Inclusion Criteria:

* infants >35 weeks of gestational age
* infants with CHD
* İnfants fed with formula feeding

Exclusion Criteria:

* Major congenital abnormalities except CHD
* infants could not be fed enterally

Ages: 8 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Weight gain | 6 weeks

SECONDARY OUTCOMES:
Neurodevelopmental evaluation | 18 months
  Neurodevelopmental evaluation will be assessed by Bayley-II Scale at corrected age of 12-18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, Study Director — Sami Ulus CH
Locations (1):
- Sami Ulus CH, Ankara, Turkey (Türkiye)